CLINICAL TRIAL: NCT02406170
Title: The REPEAT Trial: Regorafenib in Combination With Paclitaxel in Advanced Oesophagogastric Carcinoma, a Phase 1b Study
Brief Title: Regorafenib in Combination With Paclitaxel in Advanced Oesophagogastric Carcinoma
Acronym: REPEAT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, Prof.Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL.51666
Record Dates: First submitted 2015-03-26; First posted 2015-04-02 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Esophageal Neoplasms; Stomach Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Neoplasm Metastasis | interventions — regorafenib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib+Paclitaxel (Experimental): Regorafenib tolerability will be tested in a dose escalation scheme with a cytotoxic backbone of paclitaxel 80mg/m2.
  Interventions: Drug: Regorafenib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Regorafenib — The dose of regorafenib will be escalated in fixed increments to establish the maximum tolerated dose (MTD) from day 1-21 against a cytotoxic backbone of paclitaxel 80mg/m2 on days 1, 8 and 15 of a 28 day cycle
  Other Names: dose escalation scheme
Drug: Paclitaxel — Paclitaxel will be administered in combination with regorafenib to serve as a cytotoxic backbone, it will be given in a dose of 80mg/m2 on days 1,8 and 15 of a 28 day cycle.

SUMMARY:
Patients with advanced oesophagogastric cancer (OCG) have a very poor prognosis. After progression on first line therapy, second line chemotherapy with paclitaxel and a VEGF-R2 targeting antibody has a proven benefit on survival. However, no data are available on the combination of paclitaxel with kinase inhibitors in advanced OGC. Here the investigators propose a Phase 1b study to assess the tolerability of regorafenib (an oral multi kinase inhibitor) in combination with paclitaxel and to assess the uptake of paclitaxel in OCG metastasis.

DETAILED DESCRIPTION:
Rationale:

Regorafenib is a new oral multikinase inhibitor of angiogenic, stromal and oncogenic receptor tyrosine kinases. Regorafenib demonstrated to increase the overall survival of patients with metastatic colorectal cancer and has been approved by the U.S. Food and Drug Administration (FDA), as well as by The European Medicines Agency (EMA). In a recent phase IB study the combination of regorafenib with FOLFOX or FOLFIRI was shown to be a tolerable treatment regimen as first- or second-line treatment of colorectal cancer. Unfortunately, no data are available showing the effect of regorafenib on chemotherapy uptake in metastases. Here the investigators propose a phase IB study in advanced OGC with cytotoxic treatment consisting of paclitaxel together with regorafenib, to assess the tolerability of the combination as second line therapy for metastasized OGC and to assess the effect of regorafenib on paclitaxel uptake in OGC metastases.

Primary objectives:

To assess the tolerability of regorafenib combined with paclitaxel. Secondary objectives To assess the effect of regorafenib on uptake of paclitaxel in OGC metastases. To assess the effect of regorafenib on regorafenib targets in OGC metastases and blood samples.

To assess the effect of regorafenib on paclitaxel pharmacokinetics. To obtain exploratory data on the efficacy of the combination of regorafenib with paclitaxel.

Study design:

A phase 1b study of tolerability of regorafenib in combination with paclitaxel.

Study population:

Patients with advanced oesophagogastric cancer, fit for second line treatment systemic treatment.

Intervention:

The investigators will perform a phase 1b dose finding study (phase I) and then expand the cohort for evaluating the uptake of paclitaxel in OCG metastasis.

Paclitaxel will be tested as cytotoxic backbone for combination with regorafenib in advanced OGC. Paclitaxel will be dosed 80 mg/m2 I.V. infusion on Days 1, 8, and 15 of every 28 day cycle as has been reported previously and has been used in the recent RAINBOW study (NCT01170663).

Patients will receive regorafenib daily from day 1-21 of a 28-day cycle. The first cycle starting on day 2 after the first administration of chemotherapy for pharmacodynamics/kinetic purposes.

From the second cycle onwards, regorafenib will be dosed from day 1-21. Four different dose levels will be assessed. After the maximum tolerated dose (MTD) has been defined, the corresponding patient cohort will be expanded to 33 patients to assess the effect of regorafenib on uptake of paclitaxel in OGC metastases on day 1 and 15 of the first cycle (phase II).

Rationale for the starting dose:

Paclitaxel will be dosed 80 mg/m2 I.V. infusion on Days 1, 8, and 15 of every 28 day cycle as has been reported previously and has been used in the recent RAINBOW study The first dose of Regorafenib in the escalation scheme is 80mg per os qd. In phase 1 studies the optimum dose for regorafenib monotherapy has been set at 160mg per os q.d. However, considering the potential side effects of paclitaxel in combination with regorafenib the investigators chose a starting dose of 80mg per os qd.

Dose level Paclitaxel dose Regorafenib dose Minimum number patients

-1 80mg/m3 i.v 40 mg p.o. qd

1. (starting) 80mg/m3 i.v 80 mg p.o. qd 3
2. 80mg/m3 i.v 120 mg p.o. qd 3
3. 80mg/m3 i.v 160 mg p.o. qd 3

ELIGIBILITY:
Inclusion Criteria:

* Patient must understand, be willing to give consent, and sign a written informed consent form prior to undergoing any study-specific procedure
* Male or female and ≥ 18 years of age
* Metastatic or non-resectable adeno- or squamous-cell carcinoma of the stomach or oesophagus who failed on first line cytotoxic treatment with a fluoropyrimidine and platinum compound
* Tumor accessible for repeated biopsies
* Measurable or evaluable disease
* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Have adequate bone marrow, liver function, and renal function as measured by pre-specified laboratory assessments conducted within 7 days prior to the start of study treatment
* If female and of childbearing potential, have a NEGATIVE result on a pregnancy test performed a maximum of 7 days before start of study treatment
* If female and of childbearing potential or if male, must agree to use adequate contraception based on the judgment of the investigator or a designated associate from the date on which the ICF is signed until 6 months after the last dose of study drug.

Exclusion Criteria:

* Prior treatment with regorafenib
* Contra-indications for repeated biopsies
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent
* Inadequate caloric- and/or fluid intake.
* Pre-existing motor or sensory neurotoxicity greater than WHO grade 1
* ￼Have unresolved toxicity higher than National Cancer Institute-Common Terminology for Adverse Events version 4.0 (NCI-CTCAE v 4.0) Grade 1 attributed to any prior therapy/procedure, excluding alopecia.
* Have had a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of study treatment
* If female and of childbearing potential, be engaged in breast feeding
* Be unable to swallow oral tablets
* Have congestive heart failure classified as New York Heart Association Class 2 or higher
* Have had unstable angina or new-onset angina ≤ 3 months prior to screening
* Have had a myocardial infarction ≤ 6 months prior to start of study treatment
* Have cardiac arrhythmias requiring anti-arrhythmic therapy, with the exception of beta blockers or digoxin
* Have uncontrolled hypertension despite optimal medical management
* Have pheochromocytoma
* Have had arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 3 months prior to the initiation of study treatment
* Have an ongoing infection ≥ Grade 2 (NCI-CTCAE v 4.0)
* Have a known history of human immunodeficiency virus infection
* Have either active hepatitis B or C or chronic hepatitis B or C requiring treatment
* Have a seizure disorder requiring medication
* Have currently suspected brain metastases
* Have a history of organ allograft
* Have evidence or history of any bleeding diathesis (including mild hemophilia), irrespective of severity
* Have had a hemorrhage or a bleeding event > Grade 3 ( NCI-CTCAE v 4.0) within 4 weeks prior to the start of study treatment
* Have a non-healing wound, ulcer, or bone fracture
* Have interstitial lung disease with ongoing signs and symptoms at the time informed consent is obtained
* Have any other serious illness or medical condition that could jeopardize the safety of the patient
* Have an unstable illness or medical condition that could jeopardize the safety of the patient and/or his/her compliance
* Have a substance abuse, medical, psychological, or social condition that may interfere with participation in the study or evaluation of the study results
* Have a known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs
* Have any malabsorption condition
* Using and unable to stop medication that are prohibited due to interaction
* Unwilling to stop pommelos, citrus fruit and herbal medicine inducing or inhibiting the CYP system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-04; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Toxicity graded according to NCI Common Terminology Criteria for Adverse Events Version 4.0 | 4 weeks
  graded according to NCI Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE).

SECONDARY OUTCOMES:
Paclitaxel concentration in tumor biopsy | 2 year
Composite Paclitaxel pharmacokinetics | 2 year
  Area under the plasma concentration versus time curve (AUC), Peak plasma concentration (Cmax)
Expression of regorafenib targets in tumor biopsy samples | 2 year
Progression free survival | 2 years
Overall survival | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke WM van Laarhoven, MD,PHD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Medical Oncology, Amsterdam, Netherlands

REFERENCES:
- [Derived] Stroes CI, Schokker S, Khurshed M, van der Woude SO, Mathot RA, Slingerland M, de Vos-Geelen J, Zucchetti M, Matteo C, van Dijk E, Ylstra B, Thijssen V, Derks S, Godefa T, Dijksterhuis W, Breimer GE, van Delden OM, Verhoeven RH, Meijer SL, Bijlsma MF, van Laarhoven HW. A phase Ib/II study of regorafenib and paclitaxel in patients with beyond first-line advanced esophagogastric carcinoma (REPEAT). Ther Adv Med Oncol. 2022 Jun 28;14:17588359221109196. doi: 10.1177/17588359221109196. eCollection 2022. PMID 35782751